CLINICAL TRIAL: NCT06474858
Title: A Prospective Observational Study on the Effects of Obesity on Symptoms, Health Related Quality of Life and Pulmonary Function in COPD Patients
Brief Title: Effects of Obesity on COPD
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014/113
Record Dates: First submitted 2016-06-22; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: COPD; Obesity; Chronic Obstructive Pulmonary Disease
Keywords: COPD; Obesity; Chronic Obstructive Pulmonary Disease; Dyspnea; HRQoL; Symptoms; Dynamic hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Obesity; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight: COPD patients with BMI 18.5-24.99
- Obese: COPD patients with BMI ≥ 30

SUMMARY:
The purpose of this study is to investigate whether obese COPD patients experience more or less discomfort in daily life. Furthermore the investigators will evaluate if body composition or body fat distribution has effects on symptoms and performance.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) and Obesity are two major health problems. The prevalence of both is growing and there is a complex interaction between COPD and obesity. On the one hand obesity impairs lung function, with decreasing static lung volumes being the most significant effect. On the other hand there seems a beneficial role of obesity on lung function in COPD patients. This is because obese COPD patients tend to have less hyperinflation than non-obese COPD patients . An interesting question is what the net effect of these changes in lung function is on respiratory symptoms and quality of life.

In this observational study, the investigators will compare obese and non-obese COPD patients. Pulmonary function, dyspnea and quality of life will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD by a Pulmonologist defined as an obstructive lung function test with FEV1/FVC < 0.7 and FEV1 < 80% predicted
* No exacerbation of COPD at time of inclusion
* Age > 18 years
* Able to perform lung function tests and fill in the questionnaires.

Exclusion Criteria:

* Not able to perform lung function tests or fill in the questionnaires
* Diagnosis of Asthma
* Diagnosis of neuromuscular disease
* Diagnosis of heart failure
* Treatment for lung Malignancy in the past
* Active Malignancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a diagnosis of COPD who visit a Pulmonologist at Rijnstate Hospital.
Sampling Method: Probability Sample
Enrollment: 166 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Dyspnoea - mMRC | At inclusion
  Level of dyspnoea perceived in daily life measured using the Modified Medical Research Council (mMRC) dyspnoea scale. The mMRC dyspnoea scale ranges from grade 0 to 4. Higher scores mean a worse outcome.
Dyspnoea - NCSI | At inclusion
  Level of dyspnoea perceived in daily life measured using the Nijmegen Clinical Screening Instrument (NCSI). The NCSI ranges from grade 0 to 11. Higher scores mean a worse outcome.
Change in dyspnoea | Before and after the 6 minute walking test
  Level of dyspnoea using the Borg score. The Borg score ranges from grade 0 to 10. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
6 minute walking test | At inclusion
  distance walked in 6 minutes measured in metres

CONTACTS AND LOCATIONS:
Overall Officials: Safir Zewari, MD, Principal Investigator — Rijnstate Hospital, Arnhem, The Netherlands
Locations (1):
- Department Of Pulmonology, Rijnstate Hospital, The Netherlands, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: No